CLINICAL TRIAL: NCT03502486
Title: The Effects of Acute Bouts of Moderate and Intense Exercise on Alcohol and Cocaine Craving - an fNIRS Study
Brief Title: The Effects of an Acute Bout of Exercise on Alcohol and Cocaine Craving - an fNIRS Study
Acronym: ExAlCo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Basel (Other)
Collaborators: Psychiatric Hospital of the University of Basel (Other)
Responsible Party: Principal Investigator, Flora Colledge, Postdoctoral researcher, University of Basel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UBasel
Record Dates: First submitted 2018-04-05; First posted 2018-04-18 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate exercise (Experimental): 20 minutes of cycle ergometry at 50 - 60% of heart rate max.
  Interventions: Other: Moderate exercise
- Intense Exercise (Experimental): 20 minutes of cycle ergometry at 70 - 80% of heart rate max.
  Interventions: Other: Intense exercise
- Rest (Active Comparator): 20 minutes of seated reading.
  Interventions: Other: Reading

INTERVENTIONS:
Other: Moderate exercise — 20 minutes of cycle ergometry at 50-60% of heart rate max
  Arms: Moderate exercise
Other: Intense exercise — 20 minutes of cycle ergometry at 70-80% of heart rate max
  Arms: Intense Exercise
Other: Reading — 20 minutes of seated reading
  Arms: Rest

SUMMARY:
The study is a crossover randomised controlled trial. Alcohol or cocaine dependent participants will be recruited from inpatient and outpatient psychiatric treatment centres, on the approval of their treating physician. A healthy control group will be recruited using online advertising. All participants will undergo each of three conditions in a randomised order; 1) 20 minutes of cycle ergometry at 50-60% of maximum heart rate; 2) 20 minutes of exercise at 70-80% of maximum heart rate; 3) 20 minutes of quiet reading. Immediately before and after each condition, participants will be asked to complete a computerised Stroop test, watch a film containing substance-related images, and self-report craving levels. During the Stroop test and film viewing, participants' neural activity will be measured via functional near-infrared spectroscopy

DETAILED DESCRIPTION:
The aim of this study is to examine whether, following acute exercise bouts at moderate and high intensities, reduced craving and increased inhibitory control can be observed in alcohol or cocaine dependent individuals. As the focus of this study is the potential of exercise to be integrated into treatment, individuals in treatment for their dependence, who have been abstinent for a short period, will be recruited.

ELIGIBILITY:
Inclusion Criteria:

For alcohol or cocaine dependent participants:

* meeting three or more of the DSM-IV criteria for substance dependence (as determined by treating physician);
* minimum of 20 days and maximum of 40 days abstinence from substance of dependence;
* able to understand and complete the informed consent;
* able to travel to study site independently, as confirmed by the treating psychiatrist;
* assessed for physical and mental fitness by treating physician and cleared to take part in the study;
* fewer than 3 hours of physical exercise or sport per week;

For healthy controls:

* fewer than 3 hours of physical exercise or sport per week;
* no history of problematic alcohol or illicit drug consumption.

Exclusion Criteria:

* Pregnancy
* Questionable findings during resting ECG screen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Stroop test accuracy | Change from Baseline after 20 minute acute condition
  Accuracy on Stroop test
Self-reported craving | Change from Baseline after 20 minute acute condition
  Sum score on Alcohol Craving Questionnaire Short Form (scale range 12 to 84, higher scores representing greater craving) or Cocaine Craving Questionnaire - Brief (scale range 10 to 70, higher scores representing greater craving)
Cerebral oxygenation in prefrontal cortex | Change from Baseline after 20 minute acute condition
  Functional near infrared spectroscopic imaging of hemodynamic activity in prefrontal cortex
Stroop test reaction time | Change from Baseline after 20 minute acute condition
  Reaction time on Stroop test

CONTACTS AND LOCATIONS:
Overall Officials: Flora Colledge, PhD, Principal Investigator — University of Basel
Locations (1):
- Department of Sport, Exercise and Health, University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colledge F, Ludyga S, Mucke M, Puhse U, Gerber M. The effects of an acute bout of exercise on neural activity in alcohol and cocaine craving: study protocol for a randomised controlled trial. Trials. 2018 Dec 29;19(1):713. doi: 10.1186/s13063-018-3062-0. PMID 30594237